CLINICAL TRIAL: NCT02620488
Title: A Brief Laboratory-Based Hypnosis Session for Pain in Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Lonnie Zeltzer, Distinguished Professor of Pediatrics, Anesthesiology, Psychiatry and Biobehavioral Sciences, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15-000420
Record Dates: First submitted 2015-10-05; First posted 2015-12-03 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Sickle Cell Disease
Keywords: Pain Perception; Autonomic Nervous System; Sickle Cell Disease; Hypnosis; Guided Imagery
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Healthy Control (Active Comparator): Brief guided imagery session with a trained clinician focused on relaxation and pleasant imagery.
  Interventions: Behavioral: Guided Imagery
- Sickle Cell Disease (Experimental): Brief guided imagery session with a trained clinician focused on relaxation and pleasant imagery.
  Interventions: Behavioral: Guided Imagery

INTERVENTIONS:
Behavioral: Guided Imagery — Brief guided imagery session with a trained clinician focused on relaxation and pleasant imagery.

SUMMARY:
This pilot study will assess the effects of a brief laboratory-based guided imagery procedure on responses to pain in patients with sickle cell disease (SCD) and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy control or with a diagnosis of sickle cell disease
2. Age 13 or older
3. African-American
4. Subject is able to provide informed signed consent
5. Subject is able to follow instructions

Exclusion Criteria:

1. Any known acute or chronic illness that in the judgment of the investigator, may compromise subject safety or data integrity
2. Neurologic disorders affecting sensation
3. Skin abnormality/abrasion over sites of stimulus
4. Under 13 years of age
5. Unable to follow instructions

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in heart rate variability (HRV) before, during, and after hypnosis | Beginning 15 minutes prior to hypnosis session, continuing during 15 minutes of hypnosis, Ending 15 minutes after the hypnosis session
Change in galvanic skin response (GSR) before, during, and after hypnosis | Beginning 15 minutes prior to hypnosis session, continuing during 15 minutes of hypnosis, Ending 15 minutes after the hypnosis session
Change in overall respiration rate and rate of deep breathing (sighs) before, during, and after hypnosis | Beginning 15 minutes prior to hypnosis session, continuing during 15 minutes of hypnosis, Ending 15 minutes after the hypnosis session
Change in peripheral blood flow (pulse oximetry) before, during, and after hypnosis | Beginning 15 minutes prior to hypnosis session, continuing during 15 minutes of hypnosis, Ending 15 minutes after the hypnosis session

SECONDARY OUTCOMES:
Change in pain threshold temperature | 12 minutes before beginning of hypnosis session and 1 minute after end of hypnosis session
Change in pain tolerance temperature | 9 minutes before beginning of hypnosis session and 4 minutes after end of hypnosis session
Change in heat pulse pain ratings | 5 minutes before beginning of hypnosis session and 7 minutes after end of hypnosis session

CONTACTS AND LOCATIONS:
Overall Officials: Lonnie K Zeltzer, MD, Principal Investigator — UCLA Pediatric Pain and Palliative Care Program
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States